CLINICAL TRIAL: NCT04652232
Title: Randomized, Comparative Study to Assess the Effects of Cosmetic Lotion on Telogen Effluvium in Women Compared to a Control Group
Brief Title: Efficacy Study of Cosmetic Product Against Telogen Effluvium on Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RV3466F2016362
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Telogen Effluvium
Keywords: hair shedding; visual efficacy; visual effect; phototrichogram; pull test; 60-s hair count test; globalphotographs; Women
MeSH Terms: interventions — A 200 pyrinate shampoo

STUDY DESIGN:
Intervention Model Description: A randomisation list will be established. At the randomisation visit (Baseline visit 1), the Investigator will allocate a randomisation number to each subject according to the chronological order of inclusion. According to the list, the subject will be either randomized in one group of intervention.
  The investigator will only dispense the study product to the subjects included and randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Active Comparator): This group will receive the RV3466F lotion and a neutral shampoo
  Interventions: Other: RV3466F lotion; Other: Shampoo
- Control group (Other): This group will receive a neutral shampoo
  Interventions: Other: Shampoo

INTERVENTIONS:
Other: RV3466F lotion — Code: RV3466F Formula: MF5354
  Application modalities:
  3 times per week, in the evening, on a dry scalp 10 sprays overall hair after having achieved hair rays in order that the product is in contact with the scalp. Then massage to promote penetration of the lotion. Don't rinse.
  Shampoo should be avoided within the 2 hours after application
  Arms: Treated group
Other: Shampoo — Associated neutral shampoo: Extra mild shampoo Ducray® Code: RD0057H Formula: VS4031
  Application modalities:
  as often as usual
  For the treated group only : no shampoo within the 2 hours after lotion application

SUMMARY:
Telogen effluvium (TE) is one of the most common causes of non-scarring diffuse hair loss, defined as global diminution of hair with no formation of areas completely bald.

Premature termination of anagen into catagen and telogen hair follicle is the main mechanism observed in TE. It results in increased, synchronized telogen shedding leading to a decrease in global hair density.

Acute telogen effluvium (ATE) has an abrupt onset and generalized scalp hair loss occurring 2-3 months after a triggering event, which could be unidentifiable in up to 33% cases.

The degree of effluvium depends on the severity, duration of exposure and the type of agent, that can be: emotional stress, hormonal changes in the postpartum period, high fever, surgery, surgical/accidental trauma, severe haemorrhage, chronic systemic illness, or immense psychological stress, changes in medication or crash-diets. A summer effect possibly ultraviolet (UV) light induced, manifesting itself in autumn can cause ATE. The incidence of TE is not known, although it is likely that most women will experience at least 1 episode of TE during a lifetime.

ATE can be diagnosed based on relevant medical and personal history and examination subjective complaints, clinical and physical exams or relevant investigations (hair pull test, phototrichogram, blood test…). ATE generates a lot of anxiety in the patient: significant impact on quality of life, self-esteem impairment, and stress increase. Thus, stress may act as a primary inducer; an aggravating factor or be a response to hair loss.

ATE usually remits within few months (3-4 to 6 months) in 95% of cases if the trigger is removed or treated. Complete recovery may take until 1 year. A resolving TE is characterized by the absence of hair shedding, a negative hair pull test and synchronized hair growth.

In this study, our aim is to assess the effects of the RV3466F lotion on hair growth, compared to a control group, with clinical and biometrological non- invasive methods on an adult female population with telogen effluvium.

DETAILED DESCRIPTION:
In order to evaluate the interest of the RV3466F lotion in the remission of ET, which occurs naturally when the triggering cause is stopped, ,a comparative controlled group is necessary.

Moreover, due to the type of product (lotion) and the area of application ( scalp), the parallel groups design is adapted to the study purpose.

To increase the adherence to the study protocol and to limit the negative psychological impact of hair shedding without treatment, the control group receive a neutral shampoo (extra mild shampoo).

In order to avoid a bias between groups regarding the associated products, the same shampoo is given for the two groups. It should be used at the usual frequency. The allocation of the study product is randomized.

Only women are included in the study as specified in the claim of the study product.

The study area is the whole scalp. For evaluations the scalp is divided into 4 parts: centroparietal, parietal (right/left), frontal, and occipital areas The concerned part of the scalp which is evaluated can change according to the outcome measure.

The Phototrichogram (PTG) is a painless, non-invasive and objective method, used done in 2 steps 48 hours apart to provide an accurate chronological following of hair growth on a specific scalp area . All data and images are computerized, which enables a semi-automatic quantification of hair growth variables (density, growth…). A preliminary dyeing of the hair is performed, in order to enhance the contrast between hair and scalp.

The hair pull test is a semi quantitative method usually used to diagnose ongoing hair shedding and it helps to assess severity and location of hair loss.

Global photographs help to illustrate the scalp hair coverage and the overall course of hair volume. For a better standardization of the shooting conditions, a stereotactic device is used, allowing their comparison from time to time, which is done ideally by trained people, the photographs being subsequently time blinded.

The 60 seconds hair count test is a non-invasive and painless test performed by the subject itself, on the whole scalp in order to count the total number of hairs shed during a 60 seconds combing.

The clinical study includes 9 visits:

* Visit 1 - Selection (D1)
* Visit 2 - Inclusion - 48 hours (±2h) after V1
* Visit 3 - Intermediate - 4 weeks (D29 ± 4 days)
* Visit 4 -Intermediate - 48 hours (±2h) after V3
* Visit 5 - Intermediate - 8 weeks (D57 ± 4 days)
* Visit 6 - Intermediate - 48 hours (±2h) after V5
* Visit 7- Intermediate - 12 weeks (D85 ± 4 days)
* Visit 8 - Intermediate - 16 weeks (D113± 4 days)
* Visit 9 - Study end: 48 hours (±2h) after V8

The maximal duration of participation for a subject is 119 days.

ELIGIBILITY:
Selection criteria :

Criteria related to the population:

* Woman aged between 18 and 50 years old included
* Phototype I to IV included, according to Fitzpatrick classification
* Subject having signed written informed consent for the participation in the study
* Subject affiliated to a social security system or health insurance, or is a beneficiary of either (if required by national regulation)
* Subject whose last shampoo has been done at least 2 days before the selection visit
* Use of a contraceptive method assessed as efficient by an investigator (including tubal ligation), started since at least 3 months before the selection visit, continued during the study and until after 1 month after the study end
* Subject having hair length of at least 5 cm

Criteria related to diseases and hair loss disorder:

- Subject having effluvium telogen

Non selection criteria :

Criteria related to the population:

* Pregnant or breastfeeding women or planning to being pregnant during the study
* Perimenopausal symptoms (irregular menstruations, premenstrual syndrome …) or menopausal symptoms (climacteric troubles: hot flush, headaches, tiredness, insomnia, irritability …)
* Menopause (absence of menstruations since at least 1 year) or a bilateral ovariectomy
* Subject having frizzy hair
* Subject who has forfeited her freedom by administrative or legal award or is under guardianship
* Subject who, according to the judgement of the investigator, is unlikely to be compliant during the study
* Subject unable to understand the information given (for linguistic or psychiatric reasons) and to give her consent in writing to participate
* Subject who is currently participating in any another clinical trial
* Subject who has participated in another clinical trial with hair product or treatment (local on the scalp and/or systemic) within the last 12 weeks before the selection visit

Criteria related to diseases and hair loss disorders:

- Subject who has any other hair disorder or hair disease (Ludwig II, III, AA, scarring alopecia …)

Criteria related to the population:

* Pregnant or breastfeeding women or planning to being pregnant during the study
* Perimenopausal symptoms (irregular menstruations, premenstrual syndrome …) or menopausal symptoms (climacteric troubles: hot flush, headaches, tiredness, insomnia, irritability …)
* Menopause (absence of menstruations since at least 1 year) or a bilateral ovariectomy
* Subject having frizzy hair
* Subject who has forfeited her freedom by administrative or legal award or is under guardianship
* Subject who, according to the judgement of the investigator, is unlikely to be compliant during the study
* Subject unable to understand the information given (for linguistic or psychiatric reasons) and to give her consent in writing to participate
* Subject who is currently participating in any another clinical trial
* Subject who has participated in another clinical trial with hair product or treatment (local on the scalp and/or systemic) within the last 12 weeks before the selection visit

Criteria related to diseases and hair loss disorders:

* Subject who has any other hair disorder or hair disease (Ludwig II, III, AA, scarring alopecia …)
* History or clinical signs of hyperandrogenemia (menstrual cycle >35 days and hirsutism and signs of acne)
* Inflammatory skin disease or progressive skin lesion on the scalp (psoriasis, seborrheic dermatitis, severe erythema, severe excoriation, severe sunburn, etc.).
* Neoplastic disease at any time
* History of hypersensitivity or intolerance to any of the following components applied by topical route: ethyl alcohol, components of the used hair dye, components of the RV3466F lotion
* Thyroid disorders stabilised for less than 3 months

Criteria related to treatments and products:

* Systemic treatment affecting the hair growth taken for more than 4 weeks during the last 12 weeks before the selection visit:
* Finasteride
* Dutasteride
* Retinoids
* Anti-mitotic, cytotoxic drugs other than antineoplastic
* Spironolactone, flutamide, and all androgens
* Anti-epileptic agents, interferon alpha
* Minoxidil, Aminexil applied on the scalp within the last 24 weeks before the selection visit
* Systemic or local anti hair loss treatment or product, taken or applied (cosmetic solution or capsules with vitamin B, zinc, caffeine…) within the last 4 weeks before the selection visit.
* Drugs for thyroid disorders, if non stabilized for at least 3 months,
* Iron supplement if not started for at least 3 months
* Any hair care or styling method within the last week before the selection visit (e.g. dyeing, bleaching, perm, straightening, …)
* Any hair care product applied on the scalp between the last shampoo and the selection visit (e.g. gel, hairspray, wax, foam, …) or water or brushing.
* Any food supplements for hair growth taken for more than 4 weeks during the 12 weeks before the selection visit
* Radiotherapy, chemotherapy at any time
* Scalp surgery (hair transplants, laser) within the 12 months before the selection visit

Inclusion criteria :

* Criteria related to hair loss disorder:
* Subject having a proportion of hair in telogen phase superior to 15% (determined by phototrichogram at inclusion) on the centroparietal area of the scalp
* Subject having a total hair density superior or equal to ≥ 220 hairs/ cm2 (determined by phototrichogram at inclusion) on the centroparietal area of the scalp

Non inclusion criteria :

* Criteria related to treatments and products:
* Any hair care product applied on the scalp between the selection visit and the inclusion visit (e.g. gel, hairspray, wax, foam, …) or water or brushing.
* Reaction to the used hair dye during the inclusion visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
anagen to telogen ratio | Change from baseline to 16 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp

SECONDARY OUTCOMES:
anagen to telogen ratio | 1 week, 4 weeks and 8 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp
Density of telogen hair (number of hair in telogen phase/cm²) | 1 week, 4 weeks, 8 weeks and 16 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp
Density of anagen hair (number of hair in anagen phase/cm²) | 1 week, 4 weeks, 8 weeks and 16 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp
Total hair density (number of total hairs/cm²) | 1 week; 4 weeks, 8 weeks and 16 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp
Hair thickness | 1 week, 4 weeks, 8 weeks and 16 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp
Cumulative hair thickness | 1 week, 4 weeks, 8weeks and 16 weeks after application, for each group
  From phototrichogram on the centroparietal area of the scalp
Percentage of hairs pulled out | 1 week, 4 weeks, 8 weeks 12 weeks and 16 weeks after application, for each group
  From the hair pull test on right and left bitemporal areas, frontal and occipital areas.
Total number of hairs shed | 4 weeks, 8 weeks 12 weeks and 16 weeks after application, for each group
  From the 60-s hair count test on the whole scalp
Efficacy and cosmetic acceptability questionnaire | 1 week; 4 weeks, 8 weeks and 16 weeks after application, for each group
  Self-assessment questionnaire filled by the subjects. Ad-hoc questionnaires including numerical scale from 0-10 where higher scores mean a better outcome (improvement)
Density assessment | 1 week and 16 weeks after application, for each group
  From globalphotographs of the centroparietal area with a stereotactic device, blinded and assessed by experts using a 7-points scale: Important aggravation (less dense)=-3; Moderate aggravation=-2; Mild aggravation=-1; Unchanged=0; Mild improvement=1; Moderate improvement=2; Important improvement (denser)=3

CONTACTS AND LOCATIONS:
Overall Officials: Yorik Dr DROUAULT, Principal Investigator — INTERTEK FRANCE
Locations (2):
- France (2):
  - Centre de santé SABOURAUD C.E.P.C, Paris
  - INTERTEK, Paris

IPD SHARING:
Plan to Share IPD: No